CLINICAL TRIAL: NCT03776591
Title: Open D3 Right Colectomy Compared to Laparoscopic CME Right Colectomy for Right Sided Colon Cancer; an Open Randomized Controlled Study
Brief Title: Open D3 Right Hemicolectomy Compared to Laparoscopic CME for Right Sided Colon Cancer
Acronym: D3/CME
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haraldsplass Deaconess Hospital (Other)
Collaborators: Helse-Bergen HF (Other); University of Bergen (Other)
Responsible Party: Principal Investigator, Kristin Bentung Lygre, Consultant Doctor, Haraldsplass Deaconess Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REK 2015/2396
Record Dates: First submitted 2018-12-06; First posted 2018-12-14 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Complication; Quality of Life; Surgical Procedure, Unspecified; Lymph Node Metastases; Circulating Tumor Cell
Keywords: D3 lymphadenectomy; Right-sided; Colon cancer; Complications; Circulating tumor cells; Circulating DNA (cDNA); Laparoscopy; Complete mesocolic excision
MeSH Terms: conditions — Lymphatic Metastasis; Neoplastic Cells, Circulating; Colonic Neoplasms | interventions — Conversion to Open Surgery; Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open D3 (Experimental): Right colectomy Open surgery Central lymphadenectomy and vascular ligation
  Interventions: Procedure: Open surgery; Procedure: Right colectomy; Procedure: Central lymphadenectomy and vascular ligation
- Laparoscopic CME with CVL (Active Comparator): Right colectomy Laparoscopic surgery Central lymphadenectomy and vascular ligation
  Interventions: Procedure: Right colectomy; Procedure: Laparoscopic surgery; Procedure: Central lymphadenectomy and vascular ligation

INTERVENTIONS:
Procedure: Open surgery
  Arms: Open D3
Procedure: Right colectomy
Procedure: Laparoscopic surgery
  Arms: Laparoscopic CME with CVL
Procedure: Central lymphadenectomy and vascular ligation

SUMMARY:
The primary focus in this study is to investigate and improve the surgical technique. In addition the collection of clinical data during diagnostic and follow up and the collection of tumor and blood gives us the opportunity to investigate tumor biology and its relevance in terms of determine appropriate treatment strategy both surgically and oncological and to assess and predict treatment outcome.

The aim of this study is to compare short and long-term outcomes between open D3 and laparoscopic CME (complete mesocolic excision) with CVL (central vascular ligation) right colectomy for right-sided colon cancer. Our primary hypothesis is that laparoscopic surgery improves quality of life by reducing pain, postoperative complications and thereby reduces hospital stay and convalescence. On the other hand it is to prove non-inferiority of the laparoscopic group compared to the open group by means of oncological outcome (survival, recurrence). Secondary aim is to evaluate surgical quality by comparing actual vascular stump length between the two groups by postoperative CT and compare number of lymph nodes removed with the specimen. With the use of liquid biopsy we want to detect circulating tumor DNA (ctDNA) and circulating tumor cells (CTCs) and evaluate their value as tumor markers by comparing the prognostic and predictive value. The hypothesis is that ctDNA and CTCs are more sensitive than standard parameters and imaging (CT CEA).

DETAILED DESCRIPTION:
This is a prospective, randomized, multi-center clinical study. The short term outcome, 2 and 5 year survival and mortality rates will be compared between the groups operated with open D3 resection at Haukeland University hospital and laparoscopic CME with CVL right hemicolectomy at Haraldsplass Deaconess hospital. Computer generated block randomization will be used.

All patients ≤ 85 years with tumor localized in the right colon will be considered to participate in the study. The patients will be summoned to the first consultation to the hospital they are referred to. They will be informed of the study. A patient who meets the inclusion criteria will be asked to participate in the study and sign the informed consent. A patient who accepts will be assigned a sequential participant number and then referred to open D3 or laparoscopic CME (right hemicolectomy) according to a pre-specified randomized list of treatments.

All patients referred with right sided colon cancer in the inclusion period will be registered, and the reason why some do not participate in the study will be documented. Patients who decline to participate in the study will be assigned standard treatment in the institution they are referred to.

Blood samples for analysis of ctDNA/CTCs will be collected preoperatively, 3-10th postoperative day, at 3 months and at each check the next five years at six months intervals. All sample times except the first postoperative control, correspond to the time of CEA and CT in ordinary follow-up. Proteomic technology based analysis of tumor tissue

ELIGIBILITY:
Inclusion Criteria:

* • Patients with malignant tumor of the right colon (cecum, ascending colon, right flexure and right transverse) at CT, colonoscopy.

  * Patients medically cleared by anesthesiologist for general anesthesia and oncological radical resection
  * Patients ≤ 85 years
  * Signed informed consent form

Exclusion Criteria:

* • Patients with recurrent cancer after previous surgery

  * Patients with synchronous distant metastasis
  * Patients with ongoing oncological treatment due to other cancer

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Complications | 30 days
  Surgical and general complications by Clavien-Dindo Classification og surgical complications

SECONDARY OUTCOMES:
Surgical quality vascular resection | 6 months
  Vascular stump length in mm
Surgical quality lymph nodes | 6 months
  Number of lymph nodes
Patient outcome general | 6 months
  15D Health-related quality of life (HRQoL) preoperative and at 6 months. Scale 0-1. a higher score reflects a better HRQoL
Patient outcome bowel function | 6 months
  Quality of life (LARS (low anterior resection syndrome) score preoperative and at 6 months. Scale 0-42, where 0 reflects no LARS and 30-42 major LARS.
Oncological outcome survival | 60 months
  Survival in months
Oncological outcome recurrence | 60 months
  Time to recurrence in months
Prognostic significance of ctDNA | 60 months
  copies/mL plasma or % fractional abundance (mutant/total ctDNA)
Prognostic significance of CTCs | 60 months
  CTC/ml blood

OTHER OUTCOMES:
Compare the D3 specimen with the CME specimen morphologically | 4 weeks
  West classification
Operative parameters time | 1 day
  Operating time in minutes
Operative parameters blood loss | 1 day
  Intraoperative blood loss in ml
Operative parameters bleeding | 1 day
  Incidents of bleeding from central vascular structures; yes/no
Postoperative parameters | 6 months
  Incisional hernias; yes/no
Hospitalization | 30 days
  Total length of stay, including readmissions within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Kristin B. Lygre, M.D, Study Director — Haraldsplass Deaconess Hospital
Locations (1):
- Haraldsplass, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lygre KB, Forthun RB, Hoysaeter T, Hjelle SM, Eide GE, Gjertsen BT, Pfeffer F, Hovland R. Assessment of postoperative circulating tumour DNA to predict early recurrence in patients with stage I-III right-sided colon cancer: prospective observational study. BJS Open. 2024 Jan 3;8(1):zrad146. doi: 10.1093/bjsopen/zrad146. PMID 38242575
- [Derived] Lygre KB, Eide GE, Forsmo HM, Dicko A, Storli KE, Pfeffer F. Complications after open and laparoscopic right-sided colectomy with central lymphadenectomy for colon cancer: randomized controlled trial. BJS Open. 2023 Jul 10;7(4):zrad074. doi: 10.1093/bjsopen/zrad074. PMID 37643373